CLINICAL TRIAL: NCT00243165
Title: Lifemel Honey During Adjuvant Chemotherapy for Breast Cancer Patients to Prevent Leucopenia
Brief Title: Lifemel Honey to Reduce Leucopenia During Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Zuf Globus Laboratories Ltd. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LifemelCTIL
Record Dates: First submitted 2005-10-20; First posted 2005-10-21 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2005-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; honey; myelosuppression; chemotherapy
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Behavioral: Lifemel honey intake every day

SUMMARY:
This study will include 60 patients with early breast cancer referred to receive adjuvant chemotherapy with AC ( adriamycin- cyclophosphamide) or CAF ( adriamycin- cyclophosphamide- 5- fluorouracil ) combinations. These patients will receive every day one spoon of Lifemel honey or regular honey ( double blind)- during the adjuvant chemotherapy .Every week a WBC count will be performed in order to record the influence of Lifemel on myelotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patient treated with adjuvant chemotherapy
* PS = 2 or less

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-11

PRIMARY OUTCOMES:
Prevention of myelotoxicity-every week during chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Georgeta Fried, MD, Principal Investigator — Rambam Health Care Campus